CLINICAL TRIAL: NCT06322810
Title: Comparison of Erector Spiane Plan Block (ESPB) Versus Pecto-intercostal Fascial Block(PIFB) for Analgesia and Respiratory Function Recovery in Cardiac Surgery: a Randomized Control Trial
Brief Title: ESP Versus PIFB for Analgesia in Open Cardiac Surgery: a Randomized Control Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Yi-Ting Chang, Attending Anesthesiologist, Taichung Veterans General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESP vs. PIFB
Record Dates: First submitted 2024-03-10; First posted 2024-03-21 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Analgesia
Keywords: Erector spinae plane block; Pecto-intercostal plane block; Cardiac surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (Experimental): Patients who receive erector spinae plane block(ESPB) before cardiac surgery
  Interventions: Procedure: Erector spinae plane block (ESPB)
- Group P (Active Comparator): Patients who receive Pecto-intercostal plane block(PIFB) before cardiac surgery
  Interventions: Procedure: Pecto-intercostal fascial plane blok (PIFB)

INTERVENTIONS:
Procedure: Erector spinae plane block (ESPB) — Bilateral ESP: 0.5% ropivacaine 0.3 ml per kg (ideal body weight) each side, 30 min before skin excision. After surgery, use pump to deliver an intermittent automatic bolus of 0.3 ml per kg 0.16% ropivacaine every 4 hours each side.
  Arms: Group E
Procedure: Pecto-intercostal fascial plane blok (PIFB) — Bilateral PIFB: 0.5% ropivacaine 0.3 ml per kg (ideal body weight) each side, 30 min before skin excision. After surgery, use pump to deliver an intermittent automatic bolus of 0.3 ml per kg 0.16% ropivacaine every 4 hours each side.
  Arms: Group P

SUMMARY:
This clinical trial compares analgesia efficiency and recovery outcomes between two different fascial plane block techniques (ESPB vs.PIFB) in cardiac surgery patients participant population/health conditions].

The main questions it aims to answer are:

* Does ESPB provide superior analgesia than PIFB
* Do patients who receive ESPB have better recovery outcomes

DETAILED DESCRIPTION:
Regional nerve blocks, including Pecto-intercostal block (PIFB) and Erector spinae plane block (ESPB), can provide a certain level of analgesia for thoracic and cardiac surgeries. This study focuses on patients undergoing their first conventional sternotomy for cardiac surgery. They are randomly assigned to receive either PIFB or ESPB for pain relief. Comparisons are made between the two groups for postoperative 48-hour analgesic medication requirements, static and dynamic postoperative pain scores, improvements in postoperative respiratory function, quality of life index (QoL15), and other clinically relevant prognostic indicators.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients, elective and first-time cardiac surgery patients undergoing traditional sternotomy. Procedures include coronary artery bypass surgery, valve repair or replacement surgery, atrial and ventricular septal defect repair surgery, and other open-heart surgeries.

Exclusion Criteria:

* 1. Emergency surgery 2. Anticipated combined major aortic vascular surgery 3. Already admitted to the ICU or on a ventilator before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
48hr opioid consumption | Day 2
  The primary outcome of this study was the total oral morphine equivalent (OME) dose received within 48 hours after surgery. OME was calculated using a conversion toolkit within our hospital's electronic medical record system, which standardizes opioid analgesic doses to oral morphine equivalents according to established guidelines

SECONDARY OUTCOMES:
Postoperative static pain scores-Day 1 | Day 1
  Pain score reported by patients when resting
Postoperative static pain scores-Day 2 | Day 2
  Pain score reported by patients when resting
Postoperative dynamic pain scores-Day 1 | Day 1
  Pain score reported by patients when mobilizing or deep coughing
Postoperative dynamic pain scores-Day 2 | Day 2
  Pain score reported by patients when mobilizing or deep coughing
postoperative incentive spirometry volume (ml)-Day 1 | Day 1
  daily volume of incentive spirometry
postoperative incentive spirometry volume (ml)-Day 2 | Day 2
  daily volume of incentive spirometry
postoperative incentive spirometry volume (ml)-Day 3 | Day 3
  daily volume of incentive spirometry
QoL15 (pre-op) | Day 0
  quality of life questionnaire (QoL15) the day before surgery
QoL15 (POD3) | Day 3
  quality of life questionnaire (QoL15) at postoperative day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan, Taiwan